CLINICAL TRIAL: NCT01124552
Title: A Phase 2, Double-Blind, Randomized, 4-Arm, Controlled, Multi-Center Study to Evaluate the Efficacy and Safety of a Single Dose of RT001 Topical Gel for the Treatment of Moderate to Severe Lateral Canthal Lines in Adults
Brief Title: A 4-Arm Efficacy and Safety Study of RT001 for the Treatment of Moderate to Severe Lateral Canthal Lines in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RT001-CL017LCL
Record Dates: First submitted 2010-05-06; First posted 2010-05-17 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2013-12

CONDITIONS: Lateral Canthal Lines; Crow's Feet; Facial Wrinkles
Keywords: Lateral Canthal Lines; Crow's Feet Wrinkles; Facial Wrinkles

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- RT001 Botulinum toxin Type A (Dose A) (Experimental): RT001 (Botulinum toxin Type A)
  Interventions: Drug: RT001 Botulinum toxin type A (Dose A)
- RT001 Botulinum toxin type A (Dose B) (Experimental): RT001 (Botulinum Toxin Type A)
  Interventions: Drug: RT001 Botulinum Toxin Type A (Dose B)
- Dose C (Other): Vehicle Control
  Interventions: Other: Vehicle
- Dose D (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RT001 Botulinum toxin type A (Dose A) — RT001 Botulinum Toxin Type A (Dose A)
  Arms: RT001 Botulinum toxin Type A (Dose A)
Drug: RT001 Botulinum Toxin Type A (Dose B) — RT001 Botulinum Toxin Type A (Dose B)
  Arms: RT001 Botulinum toxin type A (Dose B)
Other: Vehicle — Vehicle Control
  Arms: Dose C
Drug: Placebo — Placebo Comparator
  Arms: Dose D

SUMMARY:
The purpose of this study is to find out if an investigational drug, called RT001 Topical Gel, is safe and useful in minimizing the wrinkles between the eye and hairline called lateral canthal lines, also known as crow's feet wrinkles.

DETAILED DESCRIPTION:
RT001, a new drug, may be effective for the temporary improvement in the appearance of moderate to severe lateral canthal lines (crow's feet wrinkles) in adults. In this study, researchers want to find out if RT001 is more effective than three comparator groups by examining the effect on the improvement of crow's feet by both the patient and physician.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent including authorization to release health information
* Female or male, 18 to 65 years of age and in good general health
* Willing and able to follow study instructions and likely to complete all study requirements
* Moderate to severe lateral canthal lines (crow's feet wrinkles)

Exclusion Criteria:

* Any neurological condition that may place the subject at increased risk with exposure to Botulinum Toxin Type A, including peripheral motor neuropathic diseases such as amyotrophic lateral sclerosis and motor neuropathy, and neuromuscular junctional disorders such as Lambert-Eaton syndrome and myasthenia gravis
* Muscle weakness or paralysis, particularly in the area receiving study treatment
* Active disease or irritation at the treatment areas including the eye and the skin
* Pregnant, nursing, or planning a pregnancy during the study; or is a women of child bearing potential (WOCBP) but is not willing to use an effective method of birth control
* Previous participation in a RT001 clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Subject improvement based in investigator assessment | Week 4
  The number of subjects who show improvement based on the investigator global assessment

SECONDARY OUTCOMES:
Subject Improvement Based on investigator and patient assessments | Week 4
  The number of subjects who show improvement based on the investigator global and patient assessments

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Research Institute, LLC, Coral Gables, Florida, United States